CLINICAL TRIAL: NCT00885521
Title: Exercise Training in Patients With Non-CF Bronchiectasis - a Multi-centre Randomized Controlled Trial
Brief Title: Exercise Training in Patients With Non-cystic Fibrosis (CF) Bronchiectasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: Austin Health (Other Government); Sir Charles Gairdner Hospital (Other); Curtin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 348/08
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): 8 week, twice weekly exercise program with both endurance and upper and lower limb strength training
  Interventions: Other: Exercise
- 2 (No Intervention): No exercise, twice weekly phone calls

INTERVENTIONS:
Other: Exercise — 8 week, twice weekly exercise program with endurance and upper and lower limb strength training
  Arms: Exercise

SUMMARY:
The aim of this project is to examine the short and long term effects of an 8 week, twice weekly, outpatient exercise training program for people with bronchiectasis. Participants will be randomly allocated to undergo a supervised exercise training program at The Alfred, Austin Hospital or Sir Charles Gairdner Hospital.

The hypotheses of this study are:

1. Patients with bronchiectasis who complete an exercise program will have a higher exercise capacity and better quality of life and these improvements will be sustained for up to 12 months after completion
2. Exercise training will significantly reduce the incidence of pulmonary exacerbations, use of antibiotics and rate of hospitalisation

DETAILED DESCRIPTION:
Bronchiectasis not related to cystic fibrosis (non-CF bronchiectasis) is a chronic respiratory condition characterised by permanent dilatation of the airways arising from bronchial inflammation and infection. Predominant symptoms include daily productive cough, dyspnoea and generalised fatigue. This profile is associated with diminished health-related quality of life (HRQOL) and reduced exercise tolerance.

Available medical treatments for bronchiectasis include antibiotic and inhalation therapy. To date, there is no evidence that these treatments can reduce the exacerbation rate or modify the rate of disease progression. While international guidelines for pulmonary rehabilitation recommend the inclusion of patients with bronchiectasis, there is a deficiency in evidence supporting exercise training in this population. It is proposed that a standard exercise training program conducted according to Australian guidelines for pulmonary rehabilitation will improve both exercise capacity, quality of life and reduce the number of acute infections in both the short and long term in people with bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bronchiectasis (HRCT)
* Stable medical status for last 4 weeks
* History of 2 exacerbations in the last 2 years
* Dysnpoea on exertion (Modified Medical Research Council score >1)

Exclusion Criteria:

* Concurrent diagnosis of COPD (physician diagnosis and history of 10 pack year smoking)
* Concurrent diagnosis of asthma (history of atopic disease and evidence of bronchodilator reversibility of 12% or 200ml in FEV1 or FVC)
* Concurrent diagnosis of Interstitial lung disease
* Concurrent diagnosis of Cystic Fibrosis
* Medical condition which could place patient at risk during exercise training (angina, neurological or orthopaedic condition)
* Prior completion of pulmonary rehabilitation within the last 12 months

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Incremental Shuttle Walk Test Chronic Respiratory Disease questionnaire | July 2011

SECONDARY OUTCOMES:
6-Minute Walk Test | July 2011

CONTACTS AND LOCATIONS:
Overall Officials: Annemarie L Lee, PhD, Principal Investigator — Bayside Health
Locations (3):
- Australia (3):
  - The Alfred, Melbourne, Victoria
  - Austin Health, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia

REFERENCES:
- [Derived] Lee AL, Cecins N, Holland AE, Hill CJ, McDonald CF, Burge AT, Rautela L, Thompson PJ, Stirling RG, Jenkins S. Field Walking Tests Are Reliable and Responsive to Exercise Training in People With Non-Cystic Fibrosis Bronchiectasis. J Cardiopulm Rehabil Prev. 2015 Nov-Dec;35(6):439-45. doi: 10.1097/HCR.0000000000000130. PMID 26252343
- [Derived] Lee AL, Hill CJ, Cecins N, Jenkins S, McDonald CF, Burge AT, Rautela L, Stirling RG, Thompson PJ, Holland AE. The short and long term effects of exercise training in non-cystic fibrosis bronchiectasis--a randomised controlled trial. Respir Res. 2014 Apr 15;15(1):44. doi: 10.1186/1465-9921-15-44. PMID 24731015
- [Derived] Lee AL, Cecins N, Hill CJ, Holland AE, Rautela L, Stirling RG, Thompson PJ, McDonald CF, Jenkins S. The effects of pulmonary rehabilitation in patients with non-cystic fibrosis bronchiectasis: protocol for a randomised controlled trial. BMC Pulm Med. 2010 Feb 2;10:5. doi: 10.1186/1471-2466-10-5. PMID 20122281